CLINICAL TRIAL: NCT02031341
Title: Peripheral Insulin Uptake in Type 2 Diabetes Mellitus and in Non-Diabetic Individuals
Acronym: PEAKS
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, D van Raalte, MD PhD, Amsterdam UMC, location VUmc
Other Study IDs: KGINTDVR001
Record Dates: First submitted 2014-01-03; First posted 2014-01-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes mellitus
- Normoglycemic individuals: Control group

SUMMARY:
Impaired uptake of glucose by skeletal muscle is a key feature of type 2 diabetes mellitus. It is unclear to what extent impaired insulin uptake from capillaries into skeletal muscle interstitium plays a role in this process.

We hypothesize that impaired uptake of insulin from capillaries into skeletal muscle interstitium is involved in impaired glucose uptake by skeletal muscle in type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria for all participants:

* written informed consent
* hemodynamically stable with a systolic blood pressure > 100 mmHg
* medical need to undergo a CAG procedure as determined by cardiologist

Exclusion criteria for all participants:

* ongoing myocardial infarction as determined from elevated cardiac markers
* participation in an investigational trial within 90 days prior to present study
* donation of blood (> 100 mL) within 90 days prior to present study
* serious mental impairment or language problems i.e. preventing to understand the study protocol/aim
* Use or recent use (within 3 months of study participation) of oral glucocorticoids

Inclusion criteria for non-diabetic individuals:

* 30 years ≤ age ≤ 80 years (extremes included)
* fasting glucose level of < 7.0 mmol/L and HbA1C < 6.5% (= < 48 mmol/mol)

Exclusion criteria for non-diabetic individuals:

- known T2DM/use of glucose-lowering medication

Inclusion criteria for T2DM patients:

* 30 years ≤ age ≤ 80 years (extremes included)
* fasting glucose level of > 7.0 mmol/L, or HbA1C > 6.5 (= > 48 mmol/mol) or known T2DM

Exclusion criteria for T2DM patients:

- treatment with insulin preparations

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 subjects with T2DM and 50 nondiabetic individuals
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fore-arm insulin uptake measured as ([A]-[V]) x F in pmol/min where A = arterial insulin concentrations, V= venous insulin concentrations, F = fore arm plasma flow; | Baseline
  During a single measure (thus cross-sectional) the primary endpoint will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Kennemer Gasthuis, Haarlem, Netherlands